CLINICAL TRIAL: NCT03719287
Title: National, Cross-sectional, Multicenter Study to Estimate the Point Prevalence of Peripheral Intravenous Catheter-related Complications in Brazil: a Quality Improvement Study (PIVS)
Brief Title: Study to Estimate the Point Prevalence of Peripheral Intravenous Catheter-related Complications in Brazil
Acronym: PIVS
Status: Completed | Type: Observational
Sponsor: Solventum US LLC (Industry)
Collaborators: Eurotrials Brasil Consultores Cientificos Ltda (Industry); 3M (Industry)
Responsible Party: Sponsor
Other Study IDs: EM-05-014222
Record Dates: First submitted 2018-07-23; First posted 2018-10-25 (Actual); Results first posted 2022-08-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Infusion Site Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hospital #1: Patients who meet inclusion criteria in the first of three participating Brazil hospitals
- Hospital #2: Patients who meet inclusion criteria in the second of three participating Brazil hospitals
- Hospital #3: Patients who meet inclusion criteria in the third of the three participating Brazil hospitals

SUMMARY:
A multi-center, national prevalence study where: (1) baseline SPIVC therapy complications of hospitalized adult patients that meet the inclusion/exclusion criteria of the study and (2) the compliance of clinicians to the Hospital's evidence based practice will be measured in Brazil.

DETAILED DESCRIPTION:
At each participating research site, select nurse clinicians who are experienced or experts in short peripheral I.V. catheter (SPIVC) therapy, will audit medical records and observe the SPIVC sites of adult patients in various hospital wards until a minimum total of 300 SPIVC sites are audited among 3 Brazilian acute care hospitals. The wards audited will be selected by the Investigator and will be audited during a specified time period until at least 100 SPIVCs are audited. The time to complete the study will depend on the size of the select wards, the number of nurse auditors and the number of monitoring visits required.

There are no treatments. The short peripheral I.V. catheter-related medical devices (products) observed during the study are currently approved by Brazil regulatory agencies, purchased by the hospital and available to the clinician at the time of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject, aged 18 years or older at the time of the study's audit of the ward;
* Subject admitted into one of the wards audited at the study site;
* Subject available for observation at the time of the audit;
* Subject with at least one inserted PIVC;
* Subject that voluntarily signed and dated the informed consent form (ICF) prior to study entry, if required by the study site's Ethics Committee.

Exclusion Criteria:

* Subject under treatment at the study site's outpatient clinics;
* Subject admitted into a mental health ward, emergency ward or burn unit;
* Subject awaiting transfer to another facility.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the wards of the participating acute care hospitals that will be audited in the study. To minimize subject selection bias, all subjects will be identified and invited to participate in the study consecutively, as the auditor screens the ward on the day of the audit.
Sampling Method: Non-Probability Sample
Enrollment: 295 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Simoes Neto, MD, Principal Investigator — Centro de Pequisa Clinica Sao Lucas; Larissa S Victor, RN, Principal Investigator — Hospital Erasto Gaertner (HEG); Ariane F Machado Avelar, PhD, Principal Investigator — Federal University of São Paulo
Locations (3):
- Brazil (3):
  - Hospital Erasto Gaertner (HEG), Curitiba, Paraná
  - Centro de Pequisa Clinica Sao Lucas, Campinas, São Paulo
  - Universidade Federal de Sao Paulo, São Paulo

REFERENCES:
- [Background] PR Newswire. Global Peripheral I.V. catheter market 2014-2018.
- [Background] Rickard CM, Webster J, Wallis MC, Marsh N, McGrail MR, French V, Foster L, Gallagher P, Gowardman JR, Zhang L, McClymont A, Whitby M. Routine versus clinically indicated replacement of peripheral intravenous catheters: a randomised controlled equivalence trial. Lancet. 2012 Sep 22;380(9847):1066-74. doi: 10.1016/S0140-6736(12)61082-4. PMID 22998716
- [Background] Webster J, Clarke S, Paterson D, Hutton A, van Dyk S, Gale C, Hopkins T. Routine care of peripheral intravenous catheters versus clinically indicated replacement: randomised controlled trial. BMJ. 2008 Jul 8;337(7662):a339. doi: 10.1136/bmj.a339. PMID 18614482
- [Background] Bausone-Gazda D, Lefaiver CA, Walters SA. A randomized controlled trial to compare the complications of 2 peripheral intravenous catheter-stabilization systems. J Infus Nurs. 2010 Nov-Dec;33(6):371-84. doi: 10.1097/NAN.0b013e3181f85be2. PMID 21079465
- [Background] Martinez JA, Piazuelo M, Almela M, Blecua P, Gallardo R, Rodriguez S, Escalante Z, Robau M, Trilla A. Evaluation of add-on devices for the prevention of phlebitis and other complications associated with the use of peripheral catheters in hospitalised adults: a randomised controlled study. J Hosp Infect. 2009 Oct;73(2):135-42. doi: 10.1016/j.jhin.2009.06.031. Epub 2009 Aug 27. PMID 19712998
- [Background] Maki DG. Improving the safety of peripheral intravenous catheters. BMJ. 2008 Jul 8;337(7662):a630. doi: 10.1136/bmj.a630. PMID 18614483
- [Background] Wallis MC, McGrail M, Webster J, Marsh N, Gowardman J, Playford EG, Rickard CM. Risk factors for peripheral intravenous catheter failure: a multivariate analysis of data from a randomized controlled trial. Infect Control Hosp Epidemiol. 2014 Jan;35(1):63-8. doi: 10.1086/674398. Epub 2013 Dec 2. PMID 24334800
- [Background] Alexandrou E, Ray-Barruel G, Carr PJ, Frost S, Inwood S, Higgins N, Lin F, Alberto L, Mermel L, Rickard CM. International prevalence of the use of peripheral intravenous catheters. J Hosp Med. 2015 Aug;10(8):530-3. doi: 10.1002/jhm.2389. Epub 2015 Jun 3. PMID 26041384
- [Background] Gorski LA, Hadaway L, Hagle ME, Broadhurst D, Clare S, Kleidon T, Meyer BM, Nickel B, Rowley S, Sharpe E, Alexander M. Infusion Therapy Standards of Practice, 8th Edition. J Infus Nurs. 2021 Jan-Feb 01;44(1S Suppl 1):S1-S224. doi: 10.1097/NAN.0000000000000396. No abstract available. PMID 33394637
- [Background] Mattox EA. Complications of Peripheral Venous Access Devices: Prevention, Detection, and Recovery Strategies. Crit Care Nurse. 2017 Apr;37(2):e1-e14. doi: 10.4037/ccn2017657. PMID 28365664
- [Background] Helm RE, Klausner JD, Klemperer JD, Flint LM, Huang E. Accepted but unacceptable: peripheral IV catheter failure. J Infus Nurs. 2015 May-Jun;38(3):189-203. doi: 10.1097/NAN.0000000000000100. PMID 25871866
- [Background] Marsh N, Webster J, Flynn J, Mihala G, Hewer B, Fraser J, Rickard CM. Securement methods for peripheral venous catheters to prevent failure: a randomised controlled pilot trial. J Vasc Access. 2015 May-Jun;16(3):237-44. doi: 10.5301/jva.5000348. Epub 2015 Feb 4. PMID 25656258

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hospital #1 | Hospital #2 | Hospital #3
Started | 100 | 99 | 96
Completed | 100 | 99 | 96
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline data was not analyzed per hospital
Groups:
- Total: Total of all reporting groups
Arm/Group | Hospital #1 | Hospital #2 | Hospital #3 | Total
Number analyzed (Participants) | 100 | 99 | 96 | 295
Age, Continuous [Mean (Standard Deviation); unit: Years] | NA (NA) — The age data was not analyzed per hospital | NA (NA) — The age data was not analyzed per hospital | NA (NA) — The age data was not analyzed per hospital | 54.88 (16.62)
Sex/Gender, Customized [Number; unit: participants] — The Sex/Gender data was not analyzed per hospital
  participants
    Female Participants | NA — Sex/Gender data was not analyzed per hospital | NA — Sex/Gender data was not analyzed per hospital | NA — Sex/Gender data was not analyzed per hospital | 166
    Male Participants | NA — Sex/Gender data was not analyzed per hospital | NA — Sex/Gender data was not analyzed per hospital | NA — Sex/Gender data was not analyzed per hospital | 129
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 100 | 99 | 96 | 295

OUTCOME MEASURES:

1. Primary Outcome: Percentage of PIVCs Sites With at Least One Clinical or Mechanical Complication (PIVC-related Complications)
Description: Clinical complications are: phlebitis (grade 1-4), Hematoma, Ecchymosis, Skin injury, Local infection. Mechanical complications are: Catheter dislodgement, Occlusion, Extravasation, Infiltration (grade 1-4), Leaking at the insertion site.
  Prevalence (%) = (Number of audited PIVC sites with at least one clinical or mechanical complication ÷ Number of audited PIVC sites) x 100
Time Frame: From PIVC insertion to the audit, up to 7 days.
Measure: Number (95% Confidence Interval); unit: percentage of PIVC sites
Units Other Than Participants: PIVC sites
Arm/Group | Hospital #1 | Hospital #2 | Hospital #3
Number analyzed (Participants) | 100 | 99 | 96
Number analyzed (PIVC sites) | 100 | 100 | 100
percentage of PIVC sites | 10 [4.9 to 17.6] | 6 [2.2 to 12.6] | 7 [2.9 to 13.9]

2. Secondary Outcome: Percentage of PIVC Sites With at Least One Clinical and One Mechanical Complication (PIVC-related Clinical and Mechanical Complications).
Description: Clinical complications are: phlebitis (grade 1-4), Hematoma, Ecchymosis, Skin injury, Local infection. Mechanical complications are: Catheter dislodgement, Occlusion, Extravasation, Infiltration (grade 1-4), Leaking at the insertion site.
  Prevalence (%) = (Number of audited PIVC sites with at least one clinical and one mechanical complication ÷ Number of audited PIVC sites) x 100 PIVC sites with at least one clinical complication and one mechanical complication as well.
Time Frame: From PIVC insertion to the audit, up to 7 days.
Measure: Number (95% Confidence Interval); unit: percentage of PIVC sites
Units Other Than Participants: PIVC sites
Arm/Group | Hospital #1 | Hospital #2 | Hospital #3
Number analyzed (Participants) | 100 | 99 | 96
Number analyzed (PIVC sites) | 100 | 100 | 100
percentage of PIVC sites | 0 [0 to 0] | 0 [0 to 0] | 1.0 [0 to 5.4]

3. Secondary Outcome: Percentage of PIVC Sites With at Least One Clinical Complication
Description: Specific clinical complications are: phlebitis (grade 1 - 4), Hematoma, Ecchymosis, Skin injury, Local infection.
  Prevalence (%) = (Number of audited PIVC sites with at least one clinical complication ÷ Number of audited PIVC sites) x 100
Time Frame: From PIVC insertion to the audit, up to 7 days.
Measure: Number (95% Confidence Interval); unit: percentage of PIVC sites
Units Other Than Participants: PIVC sites
Arm/Group | Hospital #1 | Hospital #2 | Hospital #3
Number analyzed (Participants) | 100 | 99 | 96
Number analyzed (PIVC sites) | 100 | 100 | 100
percentage of PIVC sites | 7.0 [2.9 to 13.9] | 5.0 [1.6 to 11.3] | 5.0 [1.6 to 11.3]

4. Secondary Outcome: Percentage of PIVC Sites With at Least One Mechanical Complication
Description: Mechanical complications are: Catheter dislodgement, Occlusion, Extravasation, Infiltration (grade 1-4), Leaking at the insertion site.
  Prevalence (%) = (Number of audited PIVC sites with at least one mechanical complication ÷ Number of audited PIVC sites) x 100
Time Frame: From PIVC insertion to the audit, up to 7 days.
Measure: Number (95% Confidence Interval); unit: percentage of PIVC sites
Units Other Than Participants: PIVC sites
Arm/Group | Hospital #1 | Hospital #2 | Hospital #3
Number analyzed (Participants) | 100 | 99 | 96
Number analyzed (PIVC sites) | 100 | 100 | 100
percentage of PIVC sites | 3.0 [0.6 to 8.5] | 1.0 [0.0 to 5.4] | 3.0 [0.6 to 8.5]

5. Secondary Outcome: Percentage of PIVC Sites With at Least One Related Quality Issue
Description: Quality Issues are: Unstable PIVC, Blood reflux,Uncontrolled IV infusion rate,Site dressing partially detached, Site dressing totally detached (site exposed to environment), Medical tape added to dressing edges, Unclean dressing, discomfort at insertion site with and without palpation, uncovered tubing access port, lack of visibility at the PIVC site.
  Prevalence (%) = (Number of audited PIVC sites with at least one related quality issue ÷ Number of audited PIVC sites) x 100
Time Frame: From PIVC insertion to the audit, up to 7 days.
Measure: Number (95% Confidence Interval); unit: percentage of PIVC sites
Arm/Group | Hospital #1 | Hospital #2 | Hospital #3
Number analyzed (Participants) | 100 | 99 | 96
percentage of PIVC sites | 61 [50.7 to 70.6] | 91 [83.6 to 95.8] | 77 [67.5 to 84.8]

ADVERSE EVENTS:
Time Frame: From PIVC insertion to the audit, up to 7 days.
Description: The country's and/or hospital's formal AE (incident) reporting process was used to document the AE.
  PIVC-related AEs corresponding to PIVC-related complications of interest for the study (Section 10.1.2) were documented by study personnel in the corresponding Individual PIVC Questionnaire. Only these events were documented in the eCFR - there was no requirement for any additional information on AEs to be recorded.
Arm/Group | Hospital #1 | Hospital #2 | Hospital #3
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/99 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/99 | 0/96
Other Adverse Events (participants affected / at risk) | 0/100 | 0/99 | 0/96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT03719287/Prot_SAP_000.pdf